CLINICAL TRIAL: NCT05187767
Title: Impact of Circulating Tumor DNA on Early Cancer Detection and Evaluation of STAS in Patients With Ground Glass Opacities
Brief Title: Impact of ctDNA in Cancer Early Detection and STAS Evaluation in Patients With GGOs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Marco Anile, Associate Professor, University of Roma La Sapienza
Other Study IDs: GGO ctDNA
Record Dates: First submitted 2021-11-15; First posted 2022-01-12 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Lung Cancer; Spreading of Tumor; Circulating Tumor Cell
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — patients serum from peripheral blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Malignant GGOs: Patients with histologically proven malignant pulmonary ground glass opacities (GGOs)
  Interventions: Diagnostic Test: cf DNA and ct DNA
- Benign GGOs: Patients with histologically or radiologically proven benign pulmonary ground glass opacities (GGOs)
  Interventions: Diagnostic Test: cf DNA and ct DNA

INTERVENTIONS:
Diagnostic Test: cf DNA and ct DNA — Quantification of the circulating free DNA and the presence of targeted circulating tumor DNA

SUMMARY:
The aim of the study is the early and non-invasive diagnosis of lung cancer in patients with pulmonary ground glass opacity. In particular, objective of the study is to evaluate the presence or absence of circulating tumor DNA (ctDNA) on the peripheral blood of patients with evidence of ground glass opacity(GGO) at CT scan and to evaluate the role that this can play in the diagnostic / therapeutic process. The ctDNA evaluation will be performed at the first radiological finding and subsequently correlated with the malignancy of the lesion based on the radiological / histological criteria regularly used in international protocols.

Secondary objective is the correlation, in patients with malignant GGO undergoing surgical treatment, of the ctDNA presence and tumor spread through the air spaces (STAS), and its correlation with local relapses.

ELIGIBILITY:
Inclusion Criteria:

* age> 18 years
* radiological finding of pulmonary ground glass opacity
* absence of solid or haematological tumor

Exclusion Criteria:

* radio / chemotherapy treatment for at least 6 months
* patient unable to understand and express his consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with radiological finding of pulmonary ground glass opacity of unknown origin
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Quantification of cf DNA | through study completion, an average of 2 year
  Assess quantity of the circulating free DNA measured in ng/μL using Qubit 2.0
Presence of ct DNA | through study completion, an average of 2 year
  Number of participants with of circulating tumor DNA using a lung pannel for genes: EGFR, KRAS, NRAS, TP53, SKT11, DDR2, PIK3CA, FGFR3, CTNNB1, MET, BRAF, ERBB2, SMAD4, PTEN, AKT, FGFR2, ERBB4, NOTCH1, FGFR1, ALK, IDH1, HRAS, IDH2, PDGFRA, RET, ROS1

CONTACTS AND LOCATIONS:
Overall Officials: Marco Anile, MD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Thoracic Surgery Unit, Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided